CLINICAL TRIAL: NCT01186055
Title: Neural Mechanisms Underlying Smoking Relapse (Center for Interdisciplinary Research on Nicotine Addiction - CIRNA)
Brief Title: Brain Activity and Smoking Cessation
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: 811325; P50CA143187 (NIH)
Record Dates: First submitted 2010-08-19; First posted 2010-08-20 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Nicotine Dependence
Keywords: Smoking Relapse; Nicotine Abstinence
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Counseling

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. A 2ml saliva sample for DNA collection & genotyping (Oragene™).
  2. A 5ml saliva sample to assess nicotine metabolites (e.g. cotinine and 3-hydroxycotinine).
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Smoking Cessation Counseling: Individuals will receive individual and group counseling for 8 weeks (6 visits) while they quit smoking.
  Interventions: Behavioral: Smoking Cessation Counseling

INTERVENTIONS:
Behavioral: Smoking Cessation Counseling — Participants shall all receive 8 weeks (6 weeks) of group or individual counseling during their quit attempt.
  Other Names: Counseling

SUMMARY:
In the current study, the investigators propose to test: (1) whether brain activation and connectivity in a resting state, assessed by ASL perfusion MRI, BOLD fMRI, and diffusion tensor imaging (DTI) predicts smoking relapse, and (2) whether brain activation, assessed by BOLD fMRI during performance of neurobehavioral probes for executive cognitive function, stress and cue reactivity, predicts smoking relapse.

DETAILED DESCRIPTION:
Our previous work demonstrated that, among non-treatment seeking smokers, regional cerebral blood flow (rCBF) is increased following 14 hours of overnight abstinence, as compared to smoking as usual. Specifically, increased rCBF was observed in the anterior cingulate, medial and left orbitofrontal cortex. Two smoking urges items ("cravings for a cigarette" and "urges to smoke at this time") that predict relapse were strongly correlated with CBF increases in several regions that comprise the brain's reward and visual circuitry (Wang et al., 2007). In addition, two other studies by our group using BOLD fMRI showed that smokers with genotypes associated with smoking relapse exhibit a reduction in BOLD signal in the bilateral dorsolateral PFC and MF/CG during nicotine withdrawal as well as impairments in working memory at high levels of task difficulty (Loughead et al., 2009). In a follow-up experiment, it was found that the smoking cessation medication varenicline reverses this deficit (Loughead et al., in press). In the current study, we propose to extend these findings in a smoking cessation treatment population by testing: (1) whether brain activation and connectivity in a resting state, assessed by ASL perfusion MRI, BOLD fMRI, and diffusion tensor imaging (DTI) predicts smoking relapse, and (2) whether brain activation, assessed by BOLD fMRI during performance of neurobehavioral probes for executive cognitive function, stress and cue reactivity, predicts smoking relapse. Following eligibility screening (week 0), 100 treatment-seeking smokers will complete two 1.5 hour pre-quit neuroimaging assessments (one following 24 hours of overnight abstinence and the other after smoking-as-usual (weeks 1 and weeks 2-3; order counterbalanced). All will receive standardized behavioral smoking cessation counseling (week 4) to prepare for a scheduled quit attempt (week 5). They will make brief visits to the Center (weeks 5, 6, 7, 8 & 9) to receive booster counseling and assess smoking status. The primary endpoints for assessing quitting success are: 8 weeks post-target quit date (week 13) and 24-weeks post target quit date (week 29). At the 8-week post-target quit date all participants will be contacted for a telephone survey and those who self-report not smoking for the past 7 days will be asked to come to the Center for biochemical confirmation. Lastly, a subset of participants (15 smokers who report having been abstinent for at least the past 7 days and 15 smokers who relapsed within the first few weeks of the TQD) will be asked to complete a third MRI scan to examine changes in brain activity related to cessation. Only those participants reporting being quit at this time point will be contacted again at 24 weeks. Identification of the neural substrates of relapse following a quit attempt could inform the development of novel medications. Further, the identification of a "brain signature" that predicts relapse may allow for the use of fMRI to screen novel medications and identify those that reverse the liability profile.

ELIGIBILITY:
Inclusion Criteria:

1. Treatment-seeking smokers between the ages of 18 and 65, reporting consumption of at least 10 cigarettes per day for at least the past 6 months.
2. Capable of giving written informed consent, which includes compliance with the requirements and restrictions listed in the combined consent and HIPAA form, and are fluent, English-speaking.
3. Provide a baseline CO reading greater than 10 parts per million (ppm) at eligibility screening.
4. Women of childbearing potential must consent to use a medically accepted method of birth control (e.g., condoms and spermicide, oral contraceptive, Depo-Provera injection, contraceptive patch, tubal ligation or abstinence from sex) for the duration of the study.

Exclusion Criteria:

Smoking Behavior

1. Use of chewing tobacco, snuff, or snus.
2. Current enrollment or plans to enroll in another research or smoking cessation program in at least the next 7 months.
3. Anticipated use (within next 7 months) of other nicotine substitutes or smoking cessation treatments/ medications.
4. Provide a baseline CO reading less than or equal to 10ppm.

Alcohol/Drug Exclusion Criteria:

1. Lifetime history of substance abuse and/or currently receiving treatment for substance abuse (e.g., alcohol, opioids, cocaine, marijuana or stimulants).
2. Current alcohol consumption that exceeds greater than 25 standard drinks/week for men and greater than 20 standard drinks/week for women over the last 6 months.
3. Breath alcohol reading (BrAC) greater than or equal to 0.01 at the Eligibility Screening or any fMRI scanning session.
4. A positive urine drug screen (cocaine, opiates, benzodiazepines, tri-cyclic antidepressants, amphetamines, methamphetamines, barbiturates, methadone, and phencyclidine) at the Eligibility Screening or any fMRI scanning session.

Medication Exclusion Criteria:

Current use or recent discontinuation (within last 2-weeks) of the following psychotropic medications:

1. Antipsychotics (typical and atypical),
2. Mood-stabilizers,
3. Anti-depressants (tricyclics, SSRI's, selective and nonselective MAOIs, Wellbutrin/Zyban),
4. Anti-panic agents,
5. Anti-obsessive agents,
6. Anti-anxiety agents,
7. Prescription (e.g., Provigil, Ritalin) or over-the-counter stimulants,
8. Diet Pills/Anorectics,
9. Systemic Steroids,
10. Varenicline,
11. Daily use of prescription medications for chronic pain.

Medical Exclusion Criteria:

1. Women who are pregnant, breast-feeding or planning a pregnancy for the duration of the study.
2. History or current diagnosis of psychosis, bipolar disorder, schizophrenia, or any Axis 1 disorder as identified by the MINI (Mini International Neuropsychiatric Interview) or self reported; for major depression, only a current diagnosis will be considered ineligible.
3. History or current diagnosis of Attention-Deficit Hyperactivity Disorder (ADHD).
4. History of epilepsy or a seizure disorder.
5. Low or borderline intellectual functioning - determined by receiving a score of less than 90 on the Shipley Institute of Living Scale (SILS) which correlates with the Wechsler Adult Intelligence Scale-Revised (WAIS-R) Estimated IQ Test (administered at the eligibility screening visit).

fMRI-Related Exclusion Criteria:

1. Participation in study #810493 or #809858 within the last 6 months.
2. History of claustrophobia.
3. Being left-handed.
4. Color blindness.
5. Lifetime history of stroke.
6. Any impairment preventing participants from using the response pad necessary for the cognitive testing.
7. Having a cochlear implant or wearing bilateral hearing aids.
8. Self-reported history of head trauma, brain or spinal tumor.
9. Self-reported use of pacemakers, certain metallic implants, or presence of metal in the eye.
10. Circumstances or conditions that may interfere with magnetic resonance imaging (MRI).
11. Self-reported history of gunshot wounds.
12. Weight greater than 250lbs at any session.

General Exclusion:

1. Participation (within the last 6 months) in other studies at our center involving cognitive testing (N-back, CPT or Go-No-Go Task).
2. Any medical condition or medication that could compromise participant safety or interfere with imaging, as determined by the Principal Investigator and/or Study Physician.
3. Inability to provide informed consent or complete any of the study tasks as determined by the Principal Investigator and/or Study Physician.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 100 treatment seeking smokers ages 18 to 65 who report smoking at least 10 cigarettes per day for at least the last 6-months.
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-04; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Association between brain activity following nicotine abstinence and quit rates after 8 weeks post-target quit date | 8 weeks
  The correlation between cerebral blood flow or BOLD signal changes and days to relapse will be examined using separate GLM analyses. For this analysis, each session's (abstinence, smoking) mean CBF (or BOLD signal) will be calculated for the ROIs. Mean values from each ROI will be used as predictors in a longitudinal logistic regression model of quitting success.

SECONDARY OUTCOMES:
Behavioral performance and BOLD signal change during neurocognitive tasks | 24 hours
  To test effect of abstinence on BOLD signal during performance of various tasks, subject-level contrast maps will be entered into a voxelwise repeated-measures session (abstinent, smoking) by ANOVA. The resulting SPM maps will be transformed to unit normal distribution SPM maps and corrected for multiple comparisons (p < 0.05) using familywise error (FWE) theory and small volume correction (SVC) procedures.
Cravings for Cigarettes | 24 hours
  During scanning sessions this assessment will be administered during the Smoking Cue task before the cue exposures, once during the task, and at the end of the task.

CONTACTS AND LOCATIONS:
Overall Officials: Caryn Lerman, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- 3535 Market Street, Suite 4100, University of Pennsylvania, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Center for Interdisciplinary Research on Nicotine Addiction — http://www.med.upenn.edu/cirna/